CLINICAL TRIAL: NCT03484338
Title: Accelerated Resolution Therapy for Treatment of Complicated Grief in Senior Adults
Brief Title: Accelerated Resolution Therapy for Complicated Grief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Kevin Kip, Distinguished Professor, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AG056584-01 (NIH)
Record Dates: First submitted 2018-03-08; First posted 2018-03-30 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Grief; Depressive Symptoms; Trauma, Psychological
MeSH Terms: conditions — Depression; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Accelerated Resolution Therapy
- Wait list controlled (Active Comparator)
  Interventions: Behavioral: Accelerated Resolution Therapy

INTERVENTIONS:
Behavioral: Accelerated Resolution Therapy — ART is an evidence-based therapy for the treatment of depressive symptoms and trauma and stress-related disorders that includes the core components of trauma-focused therapy including imaging rescripting, voluntary image replacement, guided visualization with use of eye movements, desensitization and processing of distressing memories, and in-vitro exposure to future feared triggers

SUMMARY:
This study will examine whether accelerated resolution therapy (ART) is effective for the treatment of prolonged and complicated grief and associated psychological trauma among older adult hospice caregivers who have experienced the death of an immediate family member at least 12 months ago.

DETAILED DESCRIPTION:
ART is an evidence-based therapy for the treatment of depressive symptoms and trauma and stress-related disorders that includes the core components of trauma-focused therapy including imaging rescripting, voluntary image replacement, guided visualization with use of eye movements, desensitization and processing of distressing memories, and in-vitro exposure to future feared triggers. Mental health professionals are delivering ART in clinical practice to assist with grief; however, there is a need for formal research evaluation of the effects of ART on complicated grief and psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 60 years of age or older
* previous primary caregiver of immediate family member who died after enrollment in hospice with the death occurring at least 12 months prior to enrollment
* current symptoms indicative of proposed diagnostic criteria for complicated grief disorder, as proposed by Shear et al. (2011)
* current score of >25 on the 19-item Inventory of Complicated Grief
* current symptoms indicative of significant psychological trauma, as documented by score >33on the 20-item DSM-5 PTSD checklist (PCL-5)26 or score >4 on the PDSQ PTSD subscale
* denial of suicidal ideation or intent, with no evidence of psychotic behavior

Exclusion Criteria:

* engaged in another psychotherapy regimen that could also influence symptoms of PCG - - major psychiatric disorder (e.g. bipolar disorder) deemed likely to interfere with treatment delivery
* current substance abuse dependence (alcohol and/or drug) treatment anticipated to interfere with treatment delivery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
change in complicated grief symptoms | 4 weeks, follow up at 12 weeks
  Response on the 19-item Inventory of Complicated Grief (ICF) over the course of the 4-week intervention period. Scores range from 0-76 with a score >24 indicating presence of complicated grief.
change in psychological trauma | 4 weeks, follow up at 12 weeks
  The PCL-5 (PTSD Patient Checklist)26 is a 20-item self-report instrument that will be used to assess the DSM-5 symptoms of PTSD (psychological trauma)(corresponding to criteria B-E). The total symptom severity score ranges from 0 to . A diagnostic cut-point for PTSD of 33 has been recommended. In addition, it is generally accepted that a reduction of 10 points or more on the PCL-5 is indicative of statistical and clinically meaningful improvement.
change in depressive symptoms | 4 weeks, follow up at 12 weeks
  The Center for Epidemiologic Studies Depression Scale(CES-D)37is a widely used 20-item scale that has proven useful both as a screening instrument to detect individuals at risk for depression, and to measure the symptoms of depression.

SECONDARY OUTCOMES:
change in stress response | weekly pre to post ART and over the 4 week intervention period
  For the biomarkers of sAA and IL-6, measurement will occur using the protocols listed in the Salimetrics® α-Amylase Kinetic Enzyme Assay Kit for kinetic measurement of sAA activity (Appendix B) and Salimetrics® Salivary Interleukin-6 Elisa Kit KIT (Appendix C). The unstimulated passive drool method will be used. Participants will be asked to tilt head forward, allowing the saliva to pool on the floor of the mouth, and then pass the saliva through the SalivaBio Collection Aid (SCA) into a polypropylene vial.

CONTACTS AND LOCATIONS:
Overall Officials: Harleah Buck, PhD, Principal Investigator — University of South Florida
Locations (1):
- Harleah Buck, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buck HG, Benitez B, Mason T, Hernandez D, Tofthagen C, Mogle J. Exploring the role of expectancy in older US participants' response to an accelerated resolution therapy intervention for prolonged grief disorder. Health Soc Care Community. 2022 Nov;30(6):e4191-e4198. doi: 10.1111/hsc.13813. Epub 2022 Apr 9. PMID 35396879

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03484338/Prot_SAP_000.pdf